CLINICAL TRIAL: NCT00810446
Title: DRUG USE INVESTIGATION FOR HIV INFECTION PATIENTS OF MYCOBUTIN (REGULATORY POST MARKETING COMMITMENT PLAN).
Brief Title: Safety And Efficacy Of Rifabutin In HIV Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0061007
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-06

CONDITIONS: Non-tuberculous Mycobacterial Diseases; Tuberculosis; Inhibition of Disseminated Mycobacterium Avium Complex Disease Associated With HIV Infections
MeSH Terms: conditions — Tuberculosis | interventions — Rifabutin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rifabutin: Patients administered Rifabutin.
  Interventions: Drug: rifabutin

INTERVENTIONS:
Drug: rifabutin — Mycobutin® capsules150mg depending on the Investigator prescription. Frequency and duration are according to Package Insert as follows. " 1.Tuberculosis : The usual adult dosage for oral use is 150 mg to 300 mg of rifabutin once daily.For the treatment of multiple-drug resistance tuberculosis, the usual dosage for oral use is 300 to 450 mg of rifabutin once daily.
  2.Treatment of non-tuberculous mycobacterial diseases (including MAC disease) : The usual adult dosage for oral use is 300 mg of rifabutin once daily.
  3.Inhibition of disseminated Mycobacterium avium complex (MAC) disease associated with HIV infections : The usual adult dosage for oral use is 300 mg of rifabutin once daily.".
  Other Names: Mycobutin

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Mycobutin® should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered Mycobutin® in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered Mycobutin®.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A0061007 prescribes the Mycobutin®.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0061007&StudyName=Safety%20And%20Efficacy%20Of%20Rifabutin%20In%20HIV%20Patients%0A

RESULTS

PARTICIPANT FLOW:
Groups:
- MYCOBUTIN Capsules (Rifabutin): Participants who received MYCOBUTIN Capsules as indicated in the approved local product document were observed from the start date of MYCOBUTIN Capsules administration to the completion/discontinuation. The maximum period was 8.5 years for prevention of disseminated Mycobacterium avium complex (MAC) infection in HIV and 6.5 years for treatment of tuberculosis and nontuberculous mycobacteriosis (NTM) including MAC infection. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 72 participants were registered in this study. There was no participant excluded from the baseline analysis.
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
Number analyzed (Participants) | 72
Age, Customized [Number; unit: Participants]
  <15 years | 0
  ≥15 and <65 years | 69
  ≥65 years | 3
Sex/Gender, Customized [Number; unit: Participants]
  Male | 69
  Female | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 64
  Others | 8
Diagnosis [Number; unit: Participants]
  MAC (Therapeutic) | 31
  MAC (Preventive) | 0
  Tuberculosis | 30
  NTM Infection Other Than MAC | 8
  MAC (Therapeutic) and NTM Infection Other Than MAC | 2
  Others | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Drug Reactions in This Surveillance
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to MYCOBUTIN Capsules in a participant who received MYCOBUTIN Capsules. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to MYCOBUTIN Capsules was assessed by the physician.
Time Frame: 6.5 years at maximum (therapeutic) and 8.5 years at maximum (preventive)
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received MYCOBUTIN Capsules at least once.
Measure: Number; unit: Participants
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
Number analyzed (Participants) | 72
Participants
  ADR | 16
  Serious ADR | 7

2. Primary Outcome: The Number of Participants Who Experienced an Adverse Drug Reaction Not Expected From the Local Product Document (Unknown Adverse Drug Reactions)
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to MYCOBUTIN Capsules in a participant who received MYCOBUTIN Capsules. Relatedness to MYCOBUTIN Capsules was assessed by the physician. Expectedness of the adverse drug reaction was determined according to the Japanese package insert.
Time Frame: 6.5 years at maximum (therapeutic) and 8.5 years at maximum (preventive)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
Number analyzed (Participants) | 72
Participants | 7

3. Primary Outcome: Number of Participants With Adverse Drug Reactions by Gender
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to MYCOBUTIN Capsules in a participant who received MYCOBUTIN Capsules. Relatedness to MYCOBUTIN Capsules was assessed by the physician. Participants with ADRs were counted by gender to access whether it was a risk factor for the ADR.
Time Frame: 6.5 years at maximum (therapeutic) and 8.5 years at maximum (preventive)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
Number analyzed (Participants) | 72
Participants
  Male: number analyzed (Participants) | 69
  Male | 16
  Female: number analyzed (Participants) | 3
  Female | 0

4. Primary Outcome: Number of Participants With Adverse Drug Reactions by Age
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to MYCOBUTIN Capsules in a participant who received MYCOBUTIN Capsules. Relatedness to MYCOBUTIN Capsules was assessed by the physician. Participants with ADRs were counted by age to assess whether it was a risk factor for the ADR.
Time Frame: 6.5 years at maximum (therapeutic) and 8.5 years at maximum (preventive)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
Number analyzed (Participants) | 72
Participants
  <15 years: number analyzed (Participants) | 0
  ≥15 and <65 years: number analyzed (Participants) | 69
  ≥15 and <65 years | 16
  ≥65 years: number analyzed (Participants) | 3
  ≥65 years | 0

5. Primary Outcome: Number of Participants With Adverse Drug Reactions by Diagnosis
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to MYCOBUTIN Capsules in a participant who received MYCOBUTIN Capsules. Relatedness to MYCOBUTIN Capsules was assessed by the physician. Participants with ADRs were counted by diagnosis to assess whether it was a risk factor for the ADR.
Time Frame: 6.5 years at maximum (therapeutic) and 8.5 years at maximum (preventive)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
Number analyzed (Participants) | 72
Participants
  MAC (Therapeutic): number analyzed (Participants) | 31
  MAC (Therapeutic) | 7
  MAC (Preventive): number analyzed (Participants) | 0
  Tuberculosis: number analyzed (Participants) | 30
  Tuberculosis | 8
  NTM Infections Other Than MAC: number analyzed (Participants) | 8
  NTM Infections Other Than MAC | 0
  MAC (Therapeutic) and NTM Infection Other Than MAC: number analyzed (Participants) | 2
  MAC (Therapeutic) and NTM Infection Other Than MAC | 1
  Others: number analyzed (Participants) | 1
  Others | 0

6. Primary Outcome: Clinical Response Rate (Therapeutic)
Description: Clinical response rate was defined as the percentage of participants who achieved clinical response over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Clinical efficacy of MYCOBUTIN Capsules were determined by the investigator at the final observation point based on clinical symptoms and examinations, according to the following categories: (1) markedly improved, (2) improved, (3) slightly improved (4) unchanged, (5) aggravated, or (6) indeterminable. The participants assessed as (1) markedly improved and (2) improved were considered to have achieved clinical response.
Time Frame: 6.5 years (at maximum)
Population: The effectiveness analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (overall evaluation by the physician based upon change in clinical symptoms and laboratory findings) at the final observation point. Participants assessed as "indeterminable (n=10)" at the final observation were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
Number analyzed (Participants) | 72
Percentage of Participants | 80.6 [68.63 to 89.58]

7. Primary Outcome: Clinical Response Rate (Therapeutic) by Gender
Description: Clinical response rate was defined as the percentage of participants who achieved clinical response over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Clinical efficacy of MYCOBUTIN Capsules were determined by the investigator at the final observation point based on clinical symptoms and examinations, according to the following categories: (1) markedly improved, (2) improved, (3) slightly improved (4) unchanged, (5) aggravated, or (6) indeterminable. The participants assessed as (1) markedly improved and (2) improved were considered to have achieved clinical response. Participants who achieved clinical response by gender were counted to assess whether it contributed to clinical response.
Time Frame: 6.5 years (at maximum)
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
Number analyzed (Participants) | 72
Percentage of Participants
  Male: number analyzed (Participants) | 60
  Male | 80.0
  Female: number analyzed (Participants) | 2
  Female | 100.0

8. Primary Outcome: Clinical Response Rate (Therapeutic) by Age
Description: Clinical response rate was defined as the percentage of participants who achieved clinical response over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Clinical efficacy of MYCOBUTIN Capsules were determined by the investigator at the final observation point based on clinical symptoms and examinations, according to the following categories: (1) markedly improved, (2) improved, (3) slightly improved (4) unchanged, (5) aggravated, or (6) indeterminable. The participants assessed as (1) markedly improved and (2) improved were considered to have achieved clinical response. Participants who achieved clinical response by age were counted to assess whether it contributed to clinical response.
Time Frame: 6.5 years (at maximum)
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
Number analyzed (Participants) | 72
Percentage of Participants
  <15 years: number analyzed (Participants) | 0
  ≥15 and <65 years: number analyzed (Participants) | 60
  ≥15 and <65 years | 80.0
  ≥65 years: number analyzed (Participants) | 2
  ≥65 years | 100.0

9. Primary Outcome: Clinical Response Rate (Therapeutic) by Diagnosis
Description: Clinical response rate was defined as the percentage of participants who achieved clinical response over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI. Clinical efficacy of MYCOBUTIN Capsules were determined by the investigator at the final observation point based on clinical symptoms and examinations, according to the following categories: (1) markedly improved, (2) improved, (3) slightly improved (4) unchanged, (5) aggravated, or (6) indeterminable. The participants assessed as (1) markedly improved and (2) improved were considered to have achieved clinical response. Participants who achieved clinical response by diagnosis were counted to assess whether it contributed to clinical response.
Time Frame: 6.5 years (at maximum)
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
Number analyzed (Participants) | 72
Percentage of Participants
  MAC (Therapeutic): number analyzed (Participants) | 23
  MAC (Therapeutic) | 78.3
  Tuberculosis: number analyzed (Participants) | 29
  Tuberculosis | 89.7
  NTM Infections Other Than MAC: number analyzed (Participants) | 7
  NTM Infections Other Than MAC | 57.1
  MAC (Therapeutic) and NTM Infection Other Than MAC: number analyzed (Participants) | 2
  MAC (Therapeutic) and NTM Infection Other Than MAC | 50.0
  Others: number analyzed (Participants) | 1
  Others | 100.0

ADVERSE EVENTS:
Time Frame: 6.5 years at maximum (therapeutic) and 8.5 years at maximum (preventive)
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | MYCOBUTIN Capsules (Rifabutin)
All-Cause Mortality (participants affected / at risk) | 2/72
Serious Adverse Events (participants affected / at risk) | 15/72
Other Adverse Events (participants affected / at risk) | 28/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MYCOBUTIN Capsules (Rifabutin) (N=72)
Cytomegalovirus chorioretinitis (Infections and infestations) | 3
Mycobacterium avium complex infection (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Cerebral toxoplasmosis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Atypical mycobacterial infection (Infections and infestations) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Immune reconstitution inflammatory syndrome (Immune system disorders) | 4
Irritability (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depressive symptom (Psychiatric disorders) | 1
Necrotising retinitis (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Drug resistance (General disorders) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MYCOBUTIN Capsules (Rifabutin) (N=72)
Herpes zoster (Infections and infestations) | 4
Immune reconstitution inflammatory syndrome (Immune system disorders) | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Renal impairment (Renal and urinary disorders) | 4
Blood triglycerides increased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT00810446/SAP_000.pdf
  • Study Protocol (2015-11-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT00810446/Prot_001.pdf